CLINICAL TRIAL: NCT05167825
Title: A Multicenter, Open-label, Phase III Study to Assess the Efficacy, Safety, and Pharmacokinetics of Macitentan in Japanese Pediatric Patients (>=3 Months to <15 Years) With Pulmonary Arterial Hypertension
Brief Title: A Study of Macitentan in Japanese Pediatric Participants With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109128; 67896062PAH3001 (Other: Janssen Research & Development, LLC); 2023-000984-30 (EudraCT Number)
Record Dates: First submitted 2021-11-24; First posted 2021-12-22 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Macitentan (Experimental): Participants will receive oral dose of macitentan based on age and weight through Week 52.
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan will be administered orally as a tablet.
  Other Names: OPSUMIT; ZEPENDO

SUMMARY:
The purpose of this study is to evaluate the effect of macitentan on hemodynamic measures at Week 24 in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary arterial hypertension (PAH) belonging to the nice 2013 updated classification group 1
* PAH diagnosis confirmed by historical right heart catheterization where in the absence of pulmonary vein obstruction and/or significant lung disease pulmonary artery wedge pressure (PAWP) can be replaced by left atrium pressure (LAP) or left ventricular end diastolic pressure (LVEDP) (in absence of mitral stenosis) assessed by heart catheterization
* World Health Organization (WHO) functional class (FC) I to IV
* PAH-specific treatment-naïve participants or participants on PAH-specific treatment
* A female of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) test at screening and a negative urine pregnancy test at the first administration of study intervention
* A female participant must not get pregnant and must agree not to donate eggs during the study and for a period of up to 4 weeks following the end of study

Exclusion Criteria:

* Participants with PAH due to portal hypertension, schistosomiasis, pulmonary veno-occlusive disease, and/or pulmonary capillary hemangiomatosis, and persistent pulmonary hypertension of the newborn
* Participants with the following diseases: pulmonary vein stenosis; bronchopulmonary dysplasia
* Severe hepatic impairment, example, Child-Pugh Class C, at screening
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 4 weeks after the last dose of study intervention
* Known allergies, hypersensitivity, or intolerance to macitentan or its excipients
* Participant with PAH associated with open shunts, with congenital cardiac abnormalities such as univentricular heart, with pulmonary hypertension due to lung disease, and renal dysfunction

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2025-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (11):
- Japan (11):
  - Nagano Children's Hospital, Azumino-shi
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Fukuoka Children's Hospital, Fukuoka
  - Okayama University Hospital, Okayama
  - Toho University Medical Center Omori Hospital, Ōta-ku
  - Hokkaido University Hospital, Sapporo
  - National Center for Child Health and Development, Setagaya Ku
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Osaka University Hospital, Suita-shi
  - The University of Tokyo Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7 participants were enrolled and treated in the study.
Pre-assignment Details: Results are currently reported until the primary cut-off date 24-Jul-2024. Results of remaining duration will be posted upon study completion.
Groups:
- Macitentan: Participants received macitentan 1 milligram (mg) or 2.5 mg tablets orally once daily based on age and body weight. Participants aged greater than or equal to (>=) 3 months to less than (<) 6 months received daily dose of macitentan 1 mg, >=6 months to <2 years received daily dose of macitentan 2.5 mg. For participants above 2 years (inclusive) of age, daily doses of macitentan were 3.5 mg (<15 kilograms [kg] body weight [BW]), 5 mg (>=15 kg to <25 kg BW), 7.5 mg (>=25 kg to <50 kg BW), and 10 mg (>=50 kg BW). Treatment was administered from Day 1 to Week 52.
Period: Overall Study
Arm/Group | Macitentan
Started | 7
Completed | 4
Not Completed | 3
Not completed — Ongoing | 3

BASELINE CHARACTERISTICS:
Groups:
- Macitentan: Participants aged between 3 months and 14 years, inclusive with pulmonary arterial hypertension (PAH) received macitentan 1 milligram (mg) or 2.5 mg tablets orally once daily based on age and body weight. Participants aged greater than or equal to (>=) 3 months to less than (<) 6 months received daily dose of macitentan 1 mg, >=6 months to <2 years received daily dose of macitentan 2.5 mg. For participants above 2 years (inclusive) of age, daily doses of macitentan were 3.5 mg (<15 kilograms [kg] body weight [BW]), 5 mg (>=15 kg to <25 kg BW), 7.5 mg (>=25 kg to <50 kg BW), and 10 mg (>=50 kg BW). Treatment was administered from Day 1 to Week 52 followed by 30 days follow up after end of treatment.
Arm/Group | Macitentan
Number analyzed (Participants) | 7
Age, Customized [Count of Participants; unit: Participants]
  < 2 years | 2
  >= 2 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 7

OUTCOME MEASURES:

1. Primary Outcome: Fold Change From Baseline at Week 24 in Pulmonary Vascular Resistance Index (PVRI)
Description: PVRI fold change at Week 24 was calculated as 100*(PVRI at Week 24 divided by PVRI at baseline). PVR was determined by right heart catheterization.
Time Frame: Baseline (Day 1), Week 24
Population: Efficacy analysis set included all participants who were administered at least 1 dose of macitentan.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold change (percentage)
Arm/Group | Macitentan
Number analyzed (Participants) | 7
Fold change (percentage) | 59.43 (75.1)

2. Secondary Outcome: Change From Baseline at Week 24 in Hemodynamic Variables: Pulmonary Vascular Resistance (PVR)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-03

3. Secondary Outcome: Change From Baseline in Mean Right Atrial Pressure (mRAP)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Change From Baseline at Week 24 in Hemodynamic Variables: Mean Pulmonary Arterial Pressure (mPAP)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Change From Baseline at Week 24 in Hemodynamic Variables: Cardiac Index (CI)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Change From Baseline at Week 24 in Hemodynamic Variables: Cardiac Output (CO)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Change From Baseline at Week 24 in Hemodynamic Variables: Total Pulmonary Resistance (TPR)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Change From Baseline at Week 24 in Hemodynamic Variables: Mixed Venous Oxygen Saturation (SvO2)
Time Frame: Baseline (Day 1), Week 24
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Number of Participants With Change From Baseline at Weeks 4, 8, 12, 16, 20, 24, 28, 40, and 52 in World Health Organization (WHO) Functional Class (FC)
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Number of Participants With Change From Baseline at Weeks 4, 8, 12, 16, 20, 24, 28, 40, and 52 in Panama FC
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Change From Baseline to Weeks 24 and 52 in 6-minute Walk Distance (6MWD) as Measured by the 6-minute Walk Test (6MWT)
Time Frame: Baseline (Day 1), Weeks 24 and 52
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Change From Baseline to Week 12, 24, 28, 40, and 52 in N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP)
Time Frame: Baseline (Day 1), Week 12, 24, 28, 40, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: Change From Baseline at Weeks 12, 24, and 52 in Tricuspid Annular Plane Systolic Excursion (TAPSE)
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

14. Secondary Outcome: Change From Baseline at Week 12, 24, and 52 in Left Ventricular Eccentricity Index (LVEI)
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Reporting Status: Not Posted, anticipated posting 2026-03

15. Secondary Outcome: Change From Baseline to Week 12, 24, and 52 in Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales Short Form (SF-15)
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

16. Secondary Outcome: Change From Baseline to Weeks 12, 24, and 52 in Physical Activity as Measured by Accelerometry: Number of Hours of Daytime Activity
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

17. Secondary Outcome: Change From Baseline to Weeks 12, 24, and 52 in Physical Activity as Measured by Accelerometry: Mean Count Per Minute of Daily Activity
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

18. Secondary Outcome: Change From Baseline to Weeks 12, 24, and 52 in Physical Activity as Measured by Accelerometry: Mean Daily Time Spent in Light Physical Activity
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

19. Secondary Outcome: Change From Baseline to Weeks 12, 24, and 52 in Physical Activity as Measured by Accelerometry: Mean Daily Time Spent in Moderate to Vigorous Physical Activity
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

20. Secondary Outcome: Change From Baseline to Week 24 and Week 52 in Borg Dyspnea Index
Time Frame: Baseline (Day 1), Weeks 24 and 52
Reporting Status: Not Posted, anticipated posting 2026-03

21. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: From Baseline (Day 1) up to Week 56
Reporting Status: Not Posted, anticipated posting 2026-03

22. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Time Frame: From Baseline (Day 1) up to Week 56
Reporting Status: Not Posted, anticipated posting 2026-03

23. Secondary Outcome: Number of Participants With AEs Leading to Premature Discontinuation of Macitentan
Time Frame: From Baseline (Day 1) up to Week 52
Reporting Status: Not Posted, anticipated posting 2026-03

24. Secondary Outcome: Number of Participants With AEs of Special Interest
Time Frame: From Baseline (Day 1) up to Week 56
Reporting Status: Not Posted, anticipated posting 2026-03

25. Secondary Outcome: Number of Participants With Postbaseline Markedly Abnormal Hematology Laboratory Values
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

26. Secondary Outcome: Number of Participants With Postbaseline Markedly Abnormal Clinical Chemistry Laboratory Values
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

27. Secondary Outcome: Change From Baseline in Hematology Parameters: Platelets, Leukocytes, Neutrophils Band Form, Lymphocytes, Monocytes, Eosinophils, and Basophils
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

28. Secondary Outcome: Change From Baseline in Hematology Parameters: Hematocrit
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

29. Secondary Outcome: Change From Baseline in Hematology Parameters: Hemoglobin
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

30. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocytes
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

31. Secondary Outcome: Change From Baseline in Chemistry Parameters: Sodium, Potassium, Urea Nitrogen, Glucose, and Calcium
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

32. Secondary Outcome: Change From Baseline in Chemistry Parameters: Creatinine, Bilirubin, and Direct Bilirubin
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

33. Secondary Outcome: Change From Baseline in Chemistry Parameters: Creatinine Clearance
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

34. Secondary Outcome: Change From Baseline in Chemistry Parameters: GFR From Cystatin C Adjusted for BSA
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

35. Secondary Outcome: Change From Baseline in Chemistry Parameters: Aspartate Aminotransferase, Alanine Aminotransferase, and Alkaline Phosphatase
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

36. Secondary Outcome: Change From Baseline in Vital Signs: Blood Pressure
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

37. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 40, 52
Reporting Status: Not Posted, anticipated posting 2026-03

38. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter: Heart Rate
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

39. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter: PR, QRS, QT, Corrected QT Interval-Bazett's Formula (QTcB), and Corrected QT Interval-Fridericia's Formula (QTcF)
Time Frame: Baseline (Day 1), Weeks 12, 24, and 52
Reporting Status: Not Posted, anticipated posting 2026-03

40. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: From baseline (Day 1) up to Week 56
Reporting Status: Not Posted, anticipated posting 2026-03

41. Secondary Outcome: Change From Baseline in Height
Time Frame: From baseline (Day 1) up to Week 56
Reporting Status: Not Posted, anticipated posting 2026-03

42. Secondary Outcome: Plasma Concentration of Macitentan: Participants >=2 Years Old
Time Frame: Baseline (Day 1) up to Week 12
Reporting Status: Not Posted, anticipated posting 2026-03

43. Secondary Outcome: Plasma Concentration of Aprocitentan: Participants >=2 Years Old
Time Frame: Baseline (Day 1) up to Week 12
Reporting Status: Not Posted, anticipated posting 2026-03

44. Secondary Outcome: Plasma Concentration of Macitentan: Participants <2 Years Old
Time Frame: Baseline (Day 1) up to Week 8
Reporting Status: Not Posted, anticipated posting 2026-03

45. Secondary Outcome: Plasma Concentration of Aprocitentan: Participants <2 Years Old
Time Frame: Baseline (Day 1) up to Week 8
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: All-cause mortality: From screening (Day -30) up to Week 56; Serious and Non-serious AEs: From baseline (Day 1) up to Week 56
Description: Safety analysis set included all participants who took at least 1 dose of study intervention.
Arm/Group | Macitentan
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (N=7)
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Metapneumovirus Infection (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (N=7)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Conjunctivitis Allergic (Eye disorders) | 1
Ocular Hyperaemia (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Faeces Soft (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 4
Adenovirus Infection (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 2
Conjunctivitis Bacterial (Infections and infestations) | 1
Herpes Virus Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 6
Otitis Media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia Viral (Infections and infestations) | 1
Streptococcal Infection (Infections and infestations) | 3
Upper Respiratory Tract Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 1
Crystal Urine Present (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Tongue Biting (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The interpretation of study results was limited by small sample size of only 7 participants. Study was not controlled, hence no comparison to Standard of Care (or placebo) was possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT05167825/Prot_002.pdf
  • Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT05167825/SAP_003.pdf